CLINICAL TRIAL: NCT05572242
Title: Autologous Leukocyte-platelet Rich Fibrin (L-PRF) Versus a Xenogeneic Bone Substitute Combined With a Collagen Matrix for Alveolar Ridge Preservation. A Randomized Controlled Clinical Trial
Brief Title: Leukocyte-platelet Rich Fibrin for Alveolar Ridge Preservation
Acronym: L-PRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Geistlich Pharma AG (Industry); BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Antonio Sanz, Prof., Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPI-ODO:16
Record Dates: First submitted 2022-05-03; First posted 2022-10-07 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Alveolar Ridge Enlargement
Keywords: tooth extraction; socket graft; L-PRF; xenogenic bone; dental implant

STUDY DESIGN:
Intervention Model Description: This study is a non-inferiority clinical controlled trial of parallel groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants: During the socket preservation surgery, the type of intervention will be disclosure to the surgeon. The patient will not have access to this information. Also, during the controls and following interventions (implant placement and rehabilitation), the intervention group will be masked (test or control).
  Investigator: The investigators will be always masked to the intervention group. (Only the surgeon will be able to know the treatment sequence, during the surgery) Outcomes assessor: The outcome reviewers will be blinded to the intervention. The measures of initial cbct, 4 months cbct control, and the following measurements will be always blind with respect to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- L-PRF preservation (test) (Experimental): Using L-PRF membranes inside the socket, covering with L-PRF membranes, (test group).
  Interventions: Procedure: Premolar extraction and socked preservation with L-PRF
- Xenogenic bone plus collagen membrane (control) (Active Comparator): Bio-Oss® Collagen at the bone level and application of a collagen matrix (Combi-Kit). Both materials will be used for socket preservation (control).
  Interventions: Procedure: Premolar extraction and socked preservation with Xenogenic bone and collagen membrane.

INTERVENTIONS:
Procedure: Premolar extraction and socked preservation with L-PRF — Partially edentulous patients in need of a single-tooth extraction in the premolar region[ (maxilla or mandible), with two neighboring natural teeth, will be included in the study. The tooth will be luxated first with elevators and then carefully extracted with forceps without raising a flap.
  L-PRF group will use 2-5 PRF clots, depending on the size of the socket, which will be inserted and compressed with a large plunger until they reach the alveolar crest. The site will thereafter be covered with L-PRF membranes. Then, crossed horizontal mattress suture will be placed followed by single interrupted sutures for stabilization. No efforts will be undertaken to obtain primary wound closure. The grafted socket will be left to heal for 4 months.
  After 4 months of socket preservation, a dental implant will be inserted into the socket. After 4 months of implant healing, a cad cam final restoration will be delivered. The follow-up will be up to 12 months after the final restoration.
  Arms: L-PRF preservation (test)
Procedure: Premolar extraction and socked preservation with Xenogenic bone and collagen membrane. — Partially edentulous patients in need of a single-tooth extraction in the premolar region (maxilla or mandible), with two neighboring natural teeth, will be included in the study. The tooth will be luxated first with straight and angled elevators and then carefully extracted with forceps without raising a flap.
  In the control group, the socket will be grafted with xenogeneic bone substitute material (up to the palatal/lingual bone crest) and covered with a collagen matrix. Single interrupted sutures will be placed to stabilize the collagen matrix. Sutures will be removed at 7-10 days. The grafted socket will then be left to heal for a period of 4 months.
  The xenogenic material will be Bio-Oss Collagen® and collagen matrix Bio-Gide® .
  After 4 months of socket preservation, a dental implant will be placed. After 4 months of implant healing, a cad cam final restoration will be delivered. The follow-up will be up to 12 months after the final restoration.
  Arms: Xenogenic bone plus collagen membrane (control)

SUMMARY:
After tooth extraction, there is a subsequent bone loss as a part of the natural healing of the tissue. Up to 50% of bone loss occurs during the first three months after extraction, jeopardizing a possible implant treatment. Alveolar ridge preservation techniques reduce bone loss, allowing a future implant treatment. Different bone filling materials have been used with good clinical results. The second-generation platelet concentrates (L-PRF) have recently been shown to induce bone regeneration when filling the socket after extraction, with significant biological and economic advantages. The hypothesis of this study is to test whether or not the use of L-PRF in alveolar ridge preservation results in a non-inferior horizontal radiographic change compared with the combination of a xenogeneic bone substitute with a collagen matrix.

DETAILED DESCRIPTION:
This study is a non inferiority clinical controlled trial of parallel groups. Study Intervention and Indication

After single premolar extractions in the maxilla or mandible area, patients will be randomly allocated to either one of the two treatment modalities:

* Alveolar ridge preservation using L-PRF (test)
* Alveolar ridge preservation using xenogeneic bone covered with a collagen matrix (control)

Study objectives Primary Objective The present study aims to test whether or not the use of L-PRF in alveolar ridge preservation results in non-inferior horizontal ridge width changes measured at - 1 mm below the most coronal aspect of the alveolar crest compared to the combination of a xenogeneic bone substitute material with a collagen matrix, 4 months after tooth extraction.

Clinical procedures

Extraction surgery

Partially edentulous patients in need of a single-tooth extraction in the premolar region (maxilla or mandible), with two neighboring natural teeth, will be included. All surgical procedures will be performed under local anesthesia. After disinfection of the surgical site with 0.2% chlorhexidine solution (PerioAid® Treatment, Barcelona, Spain), local anesthetics (Lidocaine HCl 2% with epinephrine 1:100,000; XXX) will be administered by infiltration at the respective buccal and lingual sites at maxilla or inferior alveolar nerve block technique on the mandible. The tooth will be luxated first with straight and angled elevators and then carefully extracted with forceps without raising a flap. After that, patients will be randomly assigned to either one of the two treatment modalities:

* Alveolar ridge preservation with leukocyte-platelet rich fibrin (L-PRF) (test)
* Alveolar ridge preservation using xenogeneic bone covered with a collagen matrix (DBBM+CM) (control)

Clinical procedures A venepuncture will be performed before any surgery (irrespective of the later randomization). Six plastic sterile 9 mL tubes without anticoagulant will be drawn with venous blood from the median basilica vein, median cubital vein, or median cephalic vein. Preparation of the L-PRF clots and membranes will be performed as previously described. In brief, within 60 seconds after the blood draws, the tubes will be centrifuged at 408 g RCF for 12 min using a tabletop centrifuge (IntraSpinTM, IntraLock®, Florida, USA). Following centrifugation, L-PRF clots will be removed from the tube, separated from the remaining red thrombus at the base with tweezers, and gently compressed into membranes using a metal rack and a metal plate.

Extraction surgery

Partially edentulous patients needing a single-tooth extraction in the premolar region (maxilla or mandible), with two neighboring natural teeth, will be included in the study. All surgical procedures will be performed under local anesthesia. After disinfection of the surgical site with 0.2% chlorhexidine solution (PerioAid® Treatment, Barcelona, Spain), local anesthetics (Lidocaine HCl 2% with epinephrine 1:100,000; XXX) will be administered by infiltration at the respective buccal and lingual sites at maxilla or inferior alveolar nerve block technique on the mandible. The tooth will be luxated first with straight and angled elevators and then carefully extracted with forceps without raising a flap. After that, patients will be randomly assigned to either one of the two treatment modalities:

* Alveolar ridge preservation with leukocyte-platelet rich fibrin (L-PRF) (test)
* Alveolar ridge preservation using xenogeneic bone covered with a collagen matrix (DBBM+CM) (control)

In group L-PRF group, 2-5 PRF clots, depending on the size of the socket, will be inserted and compressed with a large plunger until they reach the alveolar crest as previously described (Temmerman et al., 2016). The site will thereafter be covered with 2-3 L-PRF membranes. Then, crossed horizontal mattress suture will be placed, followed by single interrupted sutures for better stabilization (Vicryl 4.0 EthiconTM, Johnsson & Johnsson, New Jersey, New York, USA). No efforts will be undertaken to obtain primary wound closure. The grafted socket will be left to heal for 4 months.

In group DBBM+CM, the socket will be grafted with xenogeneic bone substitute material (up to the palatal/lingual bone crest) and covered with a collagen matrix. Single interrupted sutures (Vicryl 4.0 EthiconTM, Johnsson & Johnsson, New Jersey, New York, USA) will be placed to stabilize the collagen matrix. Sutures will be removed within 7-10 days. The grafted socket will then be left to heal for 4 months.

The xenogenic material DBBM will be Bio-Oss Collagen®, and collagen matrix Bio-Gide® both delivered as the Combi-Kit Collagen (Geistlich Pharma AG - Switzerland).

Immediately after surgery, despite the treatment group, the patient will be scanned using a CBCT (cone beam computed tomography)

Implant surgery

At 4 months, patients from both groups will be recalled for implant placement. Before the surgery, a CBCT and an impression will be taken. Moreover, clinical data will be recorded. Upon local anesthesia, a full flap will be raised, and a biopsy will be taken in the center of the implant site using a trephine drill (inner diameter 2mm). Thereafter, the implant will be placed according to the manufacturer's recommendation. A submerged healing protocol will be allowed. Final reconstructions will be inserted 4 months later.

* Type of implants: Biohorizons 3.8 * 10.5 mm as a standard implant, inserted at bone level.
* Healing mode: Submerged
* No provisional reconstruction
* Type of final reconstruction: Cad-cam screw-retained and axis screw, depending on the case.

Follow-up examinations Follow-up examinations will be performed at baseline 2 (10 days after crown insertion), 6 months, and 1 year after final restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Periodontally healthy individuals with at least 18 years of age
2. Good oral hygiene (BOP & Pl ≤ 20%)
3. Patients with a single failing premolar in the maxilla and mandible.
4. With or without buccal plate after tooth extraction (similar cases in both groups)
5. Surrounded by a mesial and distal natural tooth
6. Capability to comply with the study procedures
7. Informed Consent as documented by signature

Exclusion Criteria:

1. Pregnant or lactating women
2. Known or suspected non-compliance, drug or alcohol abuse
3. Smokers (>10 cigarettes/day)
4. Systemic or local conditions presenting a contraindication to implant treatment
5. Currently taking drugs that influence bone metabolism
6. Use of bisphosphonates in the last 4 years
7. History of malignancy, radiotherapy or chemotherapy for malignancy in the past 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Bone socket horizontal and vertical changes evaluated using cbct ((cone beam computed tomography) | first cbct immediately after socket preservation surgery, second cbct 4 months after surgery, 12 months after the final restoration of the implant.
  Cone-beam computed tomographic (CBCT) imaging will be used to assess the primary outcome (horizontal radiographic changes at -1 mm below the alveolar crest) in both groups between baseline 1 (immediately post socket preservation), visit 4 (4 months after socket preservation), and 12 months after implant rehabilitation. Linear measurements will be performed. The most apical point of the extraction socket will be defined, and two reference lines will be subsequently drawn. The vertical reference line will be drawn in the center of the extraction socket crossing the apical reference point. A horizontal reference line will be drawn perpendicular to the vertical line crossing the apical reference point. Based on these reference lines, the horizontal ridge width will then be measured at -1 mm below the alveolar crest (HW-1). The same procedure will be applied for assessing the horizontal ridge width changes will then be measured at -3 mm (HW-3) and 5- mm (HW-5) below the alveolar crest.

SECONDARY OUTCOMES:
Mucosal height | 4 months after implant insertion, at the final restoration delivery
  Mucosa height measured in millimeters from the implant platform until the mucosal margin using a North Carolina periodontal probe
Peri-implant Keratinized Mucosa | 10 days, 6, and 12 months after final restoration
  keratinized mucosal height measured in millimeters from the implant mucosal vestibular margin until the mucogingival junction using a North Carolina periodontal probe
Bleeding on probing | 10 days, 6, and 12 months after final restoration
  The presence or absence (dichotomic) of bleeding around the peri-implant sulcus after a gentle probing using a North Carolina periodontal probe
Probing depth | 10 days, 6, and 12 months after final restoration
  Probing depth of the peri-implant sulcus measured in millimeters at six points around de implant (3 points on the vestibular and 3 points on the lingual side) using a North Carolina periodontal probe
Profilometric Changes | at baseline (socket preservation), 4 months (implant insertion), 10 days and 12 months after final restoration delivery
  Profilometric changes, measured by the digitalization of stone cast obtained from de patient. The measurements will be at 1 and 3 mm below the preoperative mucosa margin.
Phenotype | 10 days, 6 and 12 months after final restoration
  Phenotype will be assessed by using a periodontal probe. If the probe results still visible after its insertion in the keratinized mucosa, the phenotype will be considered thin; if not, the phenotype will be classified as thick.
Pink esthetic score (PES) | 10 days, 6, and 12 months after final restoration
  measured at 7 sites (mesial, distal papilla, soft tissue level, soft tissue contour, bone contour, color and texture of the soft tissue) under visual examination, using 3 scores per site (0: absence, 1: partial presence, 2: full presence) with a maximum of 14 points
White esthetic score (WES) | 10 days, 6, and 12 months after final restoration
  based on tooth form, contour, color, texture, and translucence, under visual examination, using 3 scores per site (0: absence, 1: partial presence, 2: full presence) with a maximum of 14 points
Visual analog scale for pain assessment (VAS) | Pain perceived, 24 hrs after socket preservation and implant insertion (4 months).
  Ten degrees of pain are used, 0 no pain, 10 the worst pain imaginable. The patient will select a degree under his perception
Oral Health Impact Profile (OHIP-14) | at baseline, 6 and 12 months after final restoration
  self-filled questionnaire that focuses on seven dimensions of impact (functional limitation, pain, psychological discomfort, physical disability, psychological disability, social disability and handicap). Patients will be asked to respond according to frequency of impact on a 5-point Likert scale coded never (score 0), hardly ever (score 1), occasionally (score2), fairly often (score 3) and very often (score 4) using a twelve-months recall period.
  The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. Higher OHIP-14 scores indicate worse and lower scores indicate better Oral Health Related Quality of Life.
Radiographic evaluation | 10 days, 6, and 12 months after final restoration
  Intraoral calibrated X-rays images will be taken. The digitally obtained x-rays will be transferred into a software program and the pitch distance between two implant threads will be used for calibration. The marginal bone levels (MBL) will be then assessed at the mesial and distal aspects of each implant by measuring the distance between the implant shoulder and the bone crest. Thereafter, mean values will be calculated for all implants and for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Sanz, DDS, Principal Investigator — Professor
Locations (1):
- Centro de Salud, Universidad de los Andes, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No